CLINICAL TRIAL: NCT00263978
Title: Defibrotide Compassionate Use Protocol for Patients With Life Threatening Veno-Occlusive Disease of the Liver
Brief Title: Defibrotide Compassionate Use for Patients With Life Threatening Veno-Occlusive Disease of the Liver
Status: No longer available | Type: Expanded Access
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Horan, Principal Investigator, Emory University
Other Study IDs: 0966-2005
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Liver Diseases
Keywords: Venous occlusive disease; VOD
MeSH Terms: conditions — Liver Diseases | interventions — defibrotide

INTERVENTIONS:
Drug: Defibrotide

SUMMARY:
Severe veno-occlusive disease (VOD) of the liver is a life threatening complication of blood and marrow transplantation. Treatment with currently available (Food and Drug Administration [FDA] approved) agents fails in most cases. Recently conducted clinical studies indicate that patients benefit from defibrotide, a non-FDA approved agent. This protocol has been developed not with a research intent, but rather to ensure that defibrotide is used by the blood and marrow transplant programs at Children's Healthcare of Atlanta and at Emory University in a safe, effective and ethical manner.

DETAILED DESCRIPTION:
Severe veno-occlusive disease (VOD) of the liver is a life threatening complication of blood and marrow transplantation. Treatment with currently available (FDA approved) agents fails in most cases. Recently conducted clinical studies indicate that patients benefit from defibrotide, a non-FDA approved agent. This protocol has been developed not with a research intent, but rather to ensure that defibrotide is used by the blood and marrow transplant programs at Children's Healthcare of Atlanta and at Emory University in a safe, effective and ethical manner.

ELIGIBILITY:
Inclusion Criteria:

* Veno-occlusive disease of the liver

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2005-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Horan, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States